CLINICAL TRIAL: NCT01427855
Title: Saturated Fat and Protein Effects on Atherogenic Dyslipidemia
Brief Title: Dietary Protein Sources and Atherogenic Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01HL106003-01A1 (NIH); 1R01HL106003-01A1 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Disease; Dyslipidemia; Insulin Resistance; Inflammation
Keywords: Dietary Protein; Red Meat; White Meat; Vegetable Protein; Saturated Fat; LDL Subclasses; Cholesterol; Atherogenic Dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- High Saturated Fat Red Meat Diet (Experimental)
  Interventions: Other: High saturated fat red meat diet
- High Saturated Fat White Meat Diet (Experimental)
  Interventions: Other: High saturated fat white meat diet
- High Saturated Fat Non-Meat Diet (Experimental)
  Interventions: Other: High saturated fat non-meat diet
- Low Saturated Fat Red Meat Diet (Experimental)
  Interventions: Other: Low saturated fat red meat diet
- Low Saturated Fat White Meat Diet (Experimental)
  Interventions: Other: Low saturated fat white meat diet
- Low Saturated Fat Non-Meat Diet (Experimental)
  Interventions: Other: Low saturated fat non meat diet

INTERVENTIONS:
Other: High saturated fat red meat diet — 4 weeks of a high saturated fat red meat diet (38% carbohydrate; 25% protein (12% kcal from red meat protein); 37% fat (15% kcal from saturated fat))
  Arms: High Saturated Fat Red Meat Diet
Other: High saturated fat non-meat diet — 4 weeks of a high saturated fat non-meat diet (38% carbohydrate; 25% protein (16% kcal from non-meat protein); 37% fat (15% kcal from saturated fat))
  Arms: High Saturated Fat Non-Meat Diet
Other: High saturated fat white meat diet — 4 weeks of a high saturated fat white meat diet (38% carbohydrate; 25% protein (12% kcal from white meat protein); 37% fat (15% kcal from saturated fat))
  Arms: High Saturated Fat White Meat Diet
Other: Low saturated fat red meat diet — 4 weeks of a low saturated fat red meat diet (38% carbohydrate; 25% protein (12% kcal from red meat protein); 37% fat (7% kcal from saturated fat))
  Arms: Low Saturated Fat Red Meat Diet
Other: Low saturated fat white meat diet — 4 weeks of a low saturated fat white meat diet (38% carbohydrate; 25% protein (12% kcal from white meat protein); 37% fat (7% kcal from saturated fat))
  Arms: Low Saturated Fat White Meat Diet
Other: Low saturated fat non meat diet — 4 weeks of a low saturated fat non-meat diet (38% carbohydrate; 25% protein (16% kcal from non-meat protein); 37% fat (7% kcal from saturated fat))
  Arms: Low Saturated Fat Non-Meat Diet

SUMMARY:
There is growing epidemiological evidence that consumption of red meat is associated with greater incidence of Cardiovascular Disease (CVD) than either white meat or non-meat foods. Research from our group has shown that a high saturated fat (SF) diet with a moderate red meat content selectively increases intermediate density lipoproteins (IDL) and larger low density lipoproteins (LDLs), which are more weakly associated with CVD risk than smaller LDLs. In contrast, the investigators have found that with a similar intake of SF, high beef consumption results in a preferential increase in small and medium LDL particles that are strongly related to CVD. To date, no studies have directly compared the lipoprotein effects of red meat with that of other food sources of protein in the context of both high and low saturated fat intake.

The overall objective of this project is to test the hypothesis that the effects of SF on lipoprotein markers of CVD risk are influenced by sources of dietary protein. The investigators hypothesize that adverse effects of SF on plasma levels of LDL-cholesterol (C), apolipoprotein B (apo B), and atherogenic LDL particles are greater in a diet with a high content of red meat than in diets in which the major proteins are from white meat (poultry) or non-meat sources. The investigators propose a clinical trial in which 180 healthy men and women will be randomized to high SF or low SF diet groups, and within each group, consume diets with equivalent amounts of protein from red meat, white meat, and non-meat sources for 4 wks each in random order. Specifically, the investigators will test whether: (1) With high SF, the red meat diet, compared to the other protein sources, will result in higher levels of LDL-C, apoB, small and medium LDL, and total/high density lipoprotein (HDL)C; (2) With low SF, dietary protein source will not be related to any of these measurements; (3) With both the white meat and non-meat protein diets, increased LDL-C with high vs. low SF will be due primarily to increases in large LDL, whereas with red meat the additional increase in small and medium LDL will result in greater increases in plasma apoB and total LDL particle number. Aim 4 will test hypotheses that increases in small and medium LDL with high SF plus red meat are related to increased activity of hepatic lipase, a key determinant of small LDL production, and that increases in large LDL induced by high SF are related to suppression of LDL receptors. The investigators will also assess the effects of protein source and saturated fat content on markers of insulin resistance, inflammation and endothelial function.

DETAILED DESCRIPTION:
Clinic Visits:

Participants will visit the clinic a total of 11 times from screen to completion of study. This will include weekly visits with the nutritionist and 9 visits requiring blood draws (at screen and on 2 consecutive visits after each dietary period). At each visit, participants will be weighed, waist and hip circumference will be measured and blood pressure will be monitored. The total amount of blood collected during the course of the study will be 455 mL.

Screening visit (SV: 1 hour):

Recruiters will initially determine eligibility through review of a screening questionnaire and a telephone or personal interview. If a potential subject is eligible and interested, an orientation package will be mailed that will include written information about the study requirements. Interested individuals passing pre-screening will be scheduled for a screening blood draw visit to determine final eligibility. At the screening visit (SV), participants will give informed consent, review their medical history with a registered nurse, and have their blood pressure, weight, height, and waist and hip circumference measured. Thirty ml of blood will be drawn for measurement of plasma triglycerides (TG), total-C, LDL-C, HDL-C, glucose and thyroid stimulating hormone (TSH). Women of childbearing potential will be given a beta-Human Chorionic Gonadotropin (b-hCG) urine pregnancy test. Participants will be contacted within 2 weeks to notify them of their eligibility.

Nutritionist Visits (Initial: 1 hr):

Participants will meet weekly with a nutritionist to receive counseling including weight management and diet review. At these meetings, participants will receive a week's worth of frozen entrees and study foods, as well as standardized menus with check lists. During the washout period (weeks 6-8; weeks 12-14), subjects will continue to refrain from alcohol but will consume their usual home diet for 14 days.

Post-diet Visits Requiring Blood Draws (A visits: 1.5 hr, B visits: 2.5 hr):

Participants will visit the clinic on two separate days following completion of each diet to provide blood samples. Duplicate sampling reduces biological variability, and hence improves the power of the study to detect significant diet-induced changes in measurement. On the penultimate day of each diet (visits 1A, 2A, 3A, 4A) a fasting blood draw (45 mL) will be taken for plasma measurements (TG, total-C, LDL-C, HDL-C, lipoprotein subfractions, glucose, insulin, apolipoproteins AI, AII, B, and CIII, and inflammatory markers). On the last day of each dietary period (visits 1B, 2B, 3B, 4B) participants will provide a second fasting blood sample (for lipids and lipoproteins as above). Lipoprotein lipase and hepatic lipase activities will also be measured in plasma (20mL) collected 15 minutes after intravenous heparin (75 units/kg).

Clinical Procedures:

Clinical measurements: Blood pressure will be measured 3 times in a sitting position and the last 2 values averaged. Anthropometric measurements include height, weight, waist and hip circumference, and % body fat by bioimpedance (Tanita scale). Waist circumference is measured two times at the iliac crest and hip circumference is measured at the widest point of the hips.

Standard Blood sampling: Using standard blood collection procedures, blood samples will be collected from participants after a 12-14 hour fast. The blood will be collected into tubes containing the following preservative solution: 3.0 gms EDTA (dipotassium), 1.7 mg P-Pack, 0.15 gms gentamycin sulfate, 0.15 gms chloramphenicol, 5.96 mls aprotinin (Sigma A-6279), and 0.30 gms sodium azide all of which are diluted to 20mls with doubly deionized water. Plasma is separated by immediate centrifugation at 4°C. Lipid and lipoprotein measurements are performed and aliquots of plasma are frozen for future analyses.

Post-heparin Blood Sampling: A blood sample (20ml) will be drawn 15 minutes after intravenous administration of a heparin bolus (75 U/kg, see Risk section for justification) for the analysis of plasma lipase activity. Prior to administration, participants will be interviewed for family history of clotting disorders or personal contraindications including use of anticoagulants, history of bleeding or bruising abnormalities or other diseases, allergies, or recent dental work. Following administration, participants will remain in clinic for 2 hours under observation. They will also be provided with an information sheet regarding heparin and the procedure.

Measurement of endothelial function: Endothelial function will be assessed in the fasting state by finger reactive hyperemia peripheral arterial tonometry (RH-PAT, Endo-Pat2000, Itamar Medical, Israel) and expressed as RH-PAT index. Participants will rest in a supine position in a quiet, temperature-controlled room for 30 min. prior to PAT measurements and will abstain from caffeine for 6 hours and from water for 2 hours prior to the test, per manufacturer's guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old
* Non-smoking
* Agrees to abstain from alcohol and dietary supplements during the study
* Willing to consume all study foods as instructed

Exclusion Criteria:

* History of heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, lung disease, diabetes, Human immunodeficiency virus (HIV), or cancer (other than skin cancer) in the last 5 years
* Body mass index (BMI) > 35 kg/m2 or < 20 kg/m2
* Not weight stable
* Abnormal thyroid stimulating hormone
* Blood pressure > 150/90
* Fasting blood sugar >126 mg/dl
* Fasting triglyceride levels >500 mg/dl
* Total- and LDL cholesterol >95th percentile for age and sex
* Pregnant or breastfeeding
* Taking hormones or drugs known to affect lipid metabolism

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL-Cholesterol | 6 weeks, 12 weeks, 18 weeks
Change from baseline in ApoB | 6 weeks, 12 weeks, 18 weeks
Change from baseline in Small + Medium Sized LDL | 6 weeks, 12 weeks, 18 weeks
Change from baseline in Total Cholesterol/HDL Cholesterol ratio | 6 weeks, 12 weeks, 18 weeks

SECONDARY OUTCOMES:
Change from baseline in HDL-Cholesterol | 6 weeks, 12 weeks, 18 weeks
Change from baseline in non-HDLC | 6 weeks, 12 weeks, 18 weeks
Change from baseline in apoAI | 6 weeks, 12 weeks, 18 weeks
Change from baseline in apoAII | 6 weeks, 12 weeks, 18 weeks
Change from baseline in HDL2 Cholesterol | 6 weeks, 12 weeks, 18 weeks
Change from baseline in HDL3 Cholesterol | 6 weeks, 12 weeks, 18 weeks
Change from baseline in homeostasis model assessment-insulin resistance (HOMA-IR) | 6 weeks, 12 weeks, 18 weeks
Change from baseline in C-Reactive Protein | 6 weeks, 12 weeks, 18 weeks
Change from baseline in Tumor Necrosis Factor-alpha | 6 weeks, 12 weeks, 18 weeks
Change from baseline in Interleukin-6 | 6 weeks, 12 weeks, 18 weeks
Change from baseline in Monocyte Chemotactic Protein-1 (MCP-1) | 6 weeks, 12 weeks, 18 weeks
Change from baseline in RH-PAT index | 6 weeks, 12 weeks, 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Nathalie Bergeron, PhD, Principal Investigator — Children's Hospital Oakland Research Institiute
Locations (1):
- Cholesterol Research Center, Children's Hospital Research Institute, Berkeley, California, United States

REFERENCES:
- [Derived] Ferrell M, Bazeley P, Wang Z, Levison BS, Li XS, Jia X, Krauss RM, Knight R, Lusis AJ, Garcia-Garcia JC, Hazen SL, Tang WHW. Fecal Microbiome Composition Does Not Predict Diet-Induced TMAO Production in Healthy Adults. J Am Heart Assoc. 2021 Nov 2;10(21):e021934. doi: 10.1161/JAHA.121.021934. Epub 2021 Oct 29. PMID 34713713
- [Derived] Bergeron N, Chiu S, Williams PT, M King S, Krauss RM. Effects of red meat, white meat, and nonmeat protein sources on atherogenic lipoprotein measures in the context of low compared with high saturated fat intake: a randomized controlled trial. Am J Clin Nutr. 2019 Jul 1;110(1):24-33. doi: 10.1093/ajcn/nqz035. PMID 31161217